CLINICAL TRIAL: NCT02352298
Title: Protocol for the Evaluation of Dario™ Blood Glucose Monitor (BGMS) Performance at Elevated Altitude
Brief Title: Protocol for the Evaluation of Dario™ BGMS Performance at Elevated Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-0003
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dario Blood Glucose Monitoring System (Experimental): Blood obtained via fingerstick and blood glucose level is tested on the Dario Blood Glucose Monitoring System
  Interventions: Device: Dario Blood Glucose Monitoring System
- YSI STAT (Active Comparator): Blood obtained via fingerstick and blood glucose level is tested on the YSI STAT for comparison to the results obtained with the Dario Blood Glucose Monitoring System
  Interventions: Device: YSI Analyzer

INTERVENTIONS:
Device: Dario Blood Glucose Monitoring System — Fingerstick to obtain blood sample for analysis with the Dario BGMS
  Arms: Dario Blood Glucose Monitoring System
Device: YSI Analyzer — Fingerstick to obtain blood sample for analysis with YSI
  Arms: YSI STAT

SUMMARY:
The purpose of this study is to assess the performance of the Dario Blood Glucose Monitor (BGMS), at elevated altitudes, by obtaining whole blood fingerstick samples from individuals and analyzing the blood on the Dario Blood Glucose Monitor (BGMS) and comparing the readings to readings obtained from the YSI 2300 STAT Plus glucose analyzer.

DETAILED DESCRIPTION:
The study will be performed with 50 fresh capillary blood samples, collected by fingerstick using Dario single use lancet. Additional fingerstick with dedicated disposable lancets will be used to collect sufficient capillary fresh blood to be analyzed by the YSI 2300 STAT Plus analyzer. Additional fingersticks may be necessary if volume of blood from first fingerstick is insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Age of subject is 18 years or older
* Able to speak and read English

Exclusion Criteria:

* Pregnant
* Has any condition that the principal investigator believes may interfere in the subject's participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie Beatson, Study Chair — Barbara Davis Center
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 subjects - two blood glucose assessment types each (Dario vs YSI). Totaling 104 samples of blood for with 312 data points generated across 6 Dario meters and 1 YSI assessment per subject (52 total YSI assessments).
Groups:
- Dario and Yellow Springs Instrument: Blood is obtained via fingerstick and blood glucose level is tested on the Dario Blood Glucose Monitoring System, blood glucose level is then also analyzed on the Yellow Springs Instrument for comparison.
Period: Overall Study
Arm/Group | Dario and Yellow Springs Instrument
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dario and Yellow Springs Instrument: Blood obtained via fingerstick and blood glucose level is tested on the Dario Blood Glucose Monitoring System and the Yellow Springs Instrument for comparison.
Arm/Group | Dario and Yellow Springs Instrument
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 41.44 [20 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Dario Blood Glucose Monitoring System Accuracy at High Altitude (ISO 15197:2003)
Description: Accuracy of Dario Blood Glucose Monitoring System when compared to Yellow Springs Instrument 2300 reference method at 10,152 feet above sea level. Acceptance criteria set per (International Organization for Standardization) ISO 15197:2003. Greater than or equal to 95% of the Dario results shall fall within plus or minus 15 mg/dL of the reference method value (for glucose concentrations <75 mg/dL). For glucose concentrations greater than or equal to 75 mg/dL, the Dario results shall fall within plus or minus 20% of the reference method value.
Time Frame: 6 seconds
Measure: Number; unit: percentage of participants
Arm/Group | Dario Blood Glucose Monitoring System
Number analyzed (Participants) | 52
percentage of participants
  < 75 mg/dl Within ±5mg/dL | 28.6
  < 75 mg/dl Within ±10mg/dL | 71.4
  < 75 mg/dl Within ±15mg/dL | 100
  >= 75 mg/dl Within ±5% | 32.5
  >= 75 mg/dl Within ±10% | 60.1
  >=75 mg/dl Within ±15% | 87.6
  >=75 mg/dl Within ±20% | 99.2
  < 100 mg/dl Within ±5mg/dL | 28.8
  < 100 mg/dl Within ±10mg/dL | 61.4
  < 100 mg/dl Within ±15mg/dL | 97.7
  >=100 mg/dl Within ±5% | 35.7
  >=100 mg/dl Within ±10% | 65.5
  >=100 mg/dl Within ±15% | 95.2

ADVERSE EVENTS:
Arm/Group | Dario Blood Glucose Monitoring System | YSI STAT
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less